CLINICAL TRIAL: NCT06153264
Title: Effect of Neurodynamic Mobilization Exercises on Pain, Muscle Strength and Manual Dexterity in Multiple Sclerosis Patients
Brief Title: Neural Mobilization on Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Zekiye İpek KATIRCI KIRMACI, Asst. Prof, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ipek.kirmaci
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Strength; Neuro mobilization; pain
MeSH Terms: conditions — Multiple Sclerosis; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Upper extremity strengthening exercises will be applied 10 repetitions a day, 3 days a week for 6 weeks.
  Interventions: Other: strengthening exercises
- Study Group (Experimental): Upper extremity neurodynamic mobilization exercises and upper extremity strengthening exercises will be applied 10 repetitions a day, 3 days a week for 6 weeks.
  Interventions: Other: neurodynamic mobilization exercise; Other: strengthening exercises

INTERVENTIONS:
Other: neurodynamic mobilization exercise — Upper extremity neurodynamic mobilization exercises and upper extremity strengthening exercises will be applied 10 repetitions a day, 3 days a week for 6 weeks.
  Arms: Study Group
Other: strengthening exercises — upper extremity strengthening exercises will be applied 10 repetitions a day, 3 days a week for 6 weeks

SUMMARY:
Current treatments for pain in MS patients include the use of non-pharmacological interventions such as electrotherapy and exercise, as well as pharmacological treatments. Neurodynamic mobilization exercises are an intervention that aims to restore homeostasis in and around the nervous system by activating the nervous system itself or the structures surrounding the nervous system. Neurodynamic mobilization facilitates movement between neural structures and their environment through manual techniques and exercise. Human and animal studies reveal that neurodynamic mobilization reduces intraneural edema, improves intraneural fluid distribution, reduces thermal and mechanical hyperalgesia, and reverses increased immune responses following a nerve injury.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic neurological disease characterized by local inflammation, gliosis and demyelination in the central nervous system (CNS). It is characterized by demyelinating plaques seen in the brain and medulla spinalis. Many different symptoms can be seen depending on the affected areas in the CNS. One of the common symptoms in these patients is pain. Approximately 50% of patients complain of pain at some point in their lives, and in 20% of them, pain is one of the initial symptoms. Pain may originate from the musculoskeletal system; It may also develop due to inflammation and upper motor neuron damage and may have a neuropathic character. As a result, pain in MS negatively affects patients' physical, emotional functions and quality of life.

Current treatments for pain in MS patients include the use of non-pharmacological interventions such as electrotherapy and exercise, as well as pharmacological treatments. Neurodynamic mobilization exercises are an intervention that aims to restore homeostasis in and around the nervous system by activating the nervous system itself or the structures surrounding the nervous system. Neurodynamic mobilization facilitates movement between neural structures and their environment through manual techniques and exercise. Human and animal studies reveal that neurodynamic mobilization reduces intraneural edema, improves intraneural fluid distribution, reduces thermal and mechanical hyperalgesia, and reverses increased immune responses following a nerve injury.

As a result of this study, it is thought that the determination of effective treatment methods for pain, which is a common symptom of MS patients, will increase the patient's muscle strength and dexterity.

The aim of the study is to examine the effects of neurodynamic mobilization exercises on pain, muscle strength and dexterity in Multiple Sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with MS according to McDonald 2010 diagnostic criteria
2. Being between the ages of 18-65
3. Volunteering to participate in the study

Exclusion Criteria:

1. Being under 18 years of age and over 65 years of age
2. Having a history of trauma within the last year
3. Having alcohol and substance addiction
4. Having diabetes mellitus
5. Having another known neurological disease
6. Being pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline and after 6 weeks
  It is a scale used to determine the severity of pain and to clinically monitor pain.0 worst score/10 best score
Leeds Assessment of Neuropathic Symptoms and Signs Scale | Baseline and after 6 weeks
  It is a multidimensional scale based on the analysis of short-term survey data that can be applied to the patient at the bedside and is especially used to differentiate between neuropathic and nociceptive pain. The scale is scored between 0 and 24 points, and a A score higher than 12 points indicates neuropathic pain.

SECONDARY OUTCOMES:
Muscle strength | Baseline and after 6 weeks
  Upper extremity muscles will be evaluated using a digital dynamometer (Knect).
Manual Ability Measure-36 | Baseline and after 6 weeks
  In this survey, in order to evaluate manual dexterity, it is questioned how difficult it is to perform 36 activities determined to represent daily living activities without the use of assistive devices. Items are rated on a 4-point Likert-type scale from 0 (almost never performed) to 4 (easy). Scores on the 36 items were summed to create a raw total score, and then the raw scores were converted to transformed manual ability measures, which range from 0 to 100
Nine hole peg test | Baseline and after 6 weeks
  It is a validated test in MS where manual dexterity is measured in seconds based on performance. A lower time is better score.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Principal Investigator — Kahramanmaras Sütçü İmam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No